CLINICAL TRIAL: NCT05551884
Title: Non-invasive Diagnosis of Portal Hypertension in Cirrhosis Based on Metabolomics Technology(CHESS2207): a Prospective, Multicenter Study
Brief Title: Non-invasive Diagnosis of Portal Hypertension in Cirrhosis Based on Metabolomics Technology
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: The Third People's Hospital of Taiyuan (Other); Lishui Country People's Hospital (Other); Shenyang Sixth People's Hospital (Other); QuFu People's Hospital (Individual); Shulan (Hangzhou) Hospital (Other)
Responsible Party: Principal Investigator, Xiaolong Qi, Prof., Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2207
Record Dates: First submitted 2022-09-20; First posted 2022-09-23 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Cirrhosis, Liver; Portal Hypertension
Keywords: Portal hypertension; Hepatic venous pressure gradient; Non-invasive diagnostics; metabolomics
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: Training cohort was set to develop the novel non-invasive model based on metabolomics technology for HVPG.
  Interventions: Procedure: Metabolites and HVPG
- Validation cohort: Validation cohort was set to validate the novel non-invasive model based on metabolomics technology for HVPG.
  Interventions: Procedure: Metabolites and HVPG

INTERVENTIONS:
Procedure: Metabolites and HVPG — HVPG measurement are performed by well-trained interventional radiologists in accordance with standard operating procedures.
  All enrolled patients were analyzed for potential differential metabolites using metabolomics.

SUMMARY:
Portal hypertension (PH) is a group of syndromes characterized by abnormal changes in the portal blood flow system, mostly caused by cirrhosis. It is an important factor affecting the clinical prognosis of cirrhotic patients, and its severity determines the occurrence and development of cirrhotic complications.

Clinically, measurement of portal venous pressure directly is highly invasive, and factors such as intra-abdominal pressure changes can interfere with the results, limiting its clinical application. Hepatic venous pressure gradient (HVPG) is the gold standard for assessing PH in cirrhosis. The normal range of HVPG is 3~5 mmHg, and HVPG ≥5 mmHg indicates the presence of PH. AASLD stated that HVPG ≥10 mmHg is defined as clinically significant portal hypertension (CSPH), and the risk of decompensation events is significantly increased at this stage. However, HVPG is an invasive test, which is unacceptable to some patients, such as being expensive, difficult to repeat, and poor patient compliance.

Non-invasive tests for PH include serological tests, anatomical imaging and combination models. Imaging evidence of portal collateral circulation or hepatic blood flow in the portal venous system based on ultrasound Doppler, CT or magnetic resonance imaging techniques can assist to diagnose PH. In addition, elastography techniques such as transient elastography, point shear wave elastography, two-dimensional shear wave elastography and magnetic resonance elastography can be used to measure liver stiffness and spleen stiffness to assess PH. Some biochemical markers are also considered as non-invasive tests for PH. However, the available biomarkers are not yet a substitute for the HVPG accurately, and therefore, there is an urgent need for the development of biomarkers associated with HVPG in clinical practice.

Metabolomics is a method to analyze the concentrated changes of endogenous small molecule metabolites under the combined effect of genetic, biological and environmental factors with the help of various high-throughput technologies. Metabolites are at the end of the biological information flow, and their changes are the ultimate expression of the information from the coordinated action of each group, objectively reflecting the overall changes of the organism. Currently, metabolomics techniques have been widely used in screening biomarkers of liver diseases. Wang et al. applied GC-TOF/MS and UPLC-QTOF/MS to study the urinary metabolomics of patients with hepatitis B cirrhosis and showed that α-hydroxymaurolate, tyrosine-betaine, 3-hydroxyisovaleric acid, knife-serine succinate, estrone and GUDCA were significantly altered in different Child-Pugh grades of cirrhosis, suggesting that these metabolites are potential biomarkers to identify different pathological stages of cirrhosis. Therefore, metabolomics is a reliable and valid tool for biomarker discovery.

In conclusion, this study analyzed significantly altered metabolites in patients with hepatitis B cirrhosis using metabolomics to explore potential differential metabolites that are highly correlated with HVPG. Further, serological biomarkers were identified as an alternative to HVPG testing through model construction and validation.

DETAILED DESCRIPTION:
Portal hypertension (PH) is a group of syndromes characterized by abnormal changes in the portal blood flow system, mostly caused by cirrhosis. It is an important factor affecting the clinical prognosis of cirrhotic patients, and its severity determines the occurrence and development of cirrhotic complications.

Clinically, measurement of portal venous pressure directly is highly invasive, and factors such as intra-abdominal pressure changes can interfere with the results, limiting its clinical application. Hepatic venous pressure gradient (HVPG) is the gold standard for assessing PH in cirrhosis. The normal range of HVPG is 3~5 mmHg, and HVPG ≥5 mmHg indicates the presence of PH. AASLD stated that HVPG ≥10 mmHg is defined as clinically significant portal hypertension (CSPH), and the risk of decompensation events is significantly increased at this stage. However, HVPG is an invasive test, which is unacceptable to some patients, such as being expensive, difficult to repeat, and poor patient compliance.

Non-invasive tests for PH include serological tests, anatomical imaging and combination models. Imaging evidence of portal collateral circulation or hepatic blood flow in the portal venous system based on ultrasound Doppler, CT or magnetic resonance imaging techniques can assist to diagnose PH. In addition, elastography techniques such as transient elastography, point shear wave elastography, two-dimensional shear wave elastography and magnetic resonance elastography can be used to measure liver stiffness and spleen stiffness to assess PH. Some biochemical markers are also considered as non-invasive tests for PH. A study by Buck's team showed that serum inflammatory markers in cirrhotic patients were highly correlated with HVPG. Liver fibrosis index has been proposed for the grading and identification of fibrosis with moderate accuracy. Bone bridging protein levels were also correlated with the degree of liver fibrosis and CSPH. Overall, non-invasive serological markers have great potential in assessing PH. However, the available biomarkers are not yet a substitute for the HVPG accurately, and therefore, there is an urgent need for the development of biomarkers associated with HVPG in clinical practice.

Metabolomics is a method to analyze the concentrated changes of endogenous small molecule metabolites under the combined effect of genetic, biological and environmental factors with the help of various high-throughput technologies. Metabolites are at the end of the biological information flow, and their changes are the ultimate expression of the information from the coordinated action of each group, objectively reflecting the overall changes of the organism. Currently, metabolomics techniques have been widely used in screening biomarkers of liver diseases. Wang et al. applied GC-TOF/MS and UPLC-QTOF/MS to study the urinary metabolomics of patients with hepatitis B cirrhosis and showed that α-hydroxymaurolate, tyrosine-betaine, 3-hydroxyisovaleric acid, knife-serine succinate, estrone and GUDCA were significantly altered in different Child-Pugh grades of cirrhosis, suggesting that these metabolites are potential biomarkers to identify different pathological stages of cirrhosis. Therefore, metabolomics is a reliable and valid tool for biomarker discovery.

In conclusion, this study analyzed significantly altered metabolites in patients with hepatitis B cirrhosis using metabolomics to explore potential differential metabolites that are highly correlated with HVPG. Further, serological biomarkers were identified as an alternative to HVPG testing through model construction and validation.

ELIGIBILITY:
Inclusion Criteria:

1. Case group: age 18-75 years old; patients with hepatitis B cirrhosis diagnosed by liver biopsy, or definite clinical data, or imaging findings; undergo HVPG examination; with written informed consent.
2. Control group: no liver-related diseases, matched with the case group in terms of race, age, sex, and BMI.

Exclusion Criteria:

1. Other etiologies caused cirrhosis, such as HCV, autoimmune hepatitis, alcoholic, non-alcoholic liver disease, etc;
2. Patients with severe liver failure, hepatocellular carcinoma, portal vein thrombosis.
3. Patients with recent blood transfusion due to bleeding.
4. Patients who are pregnant or lactating.
5. Patients with endocrine and metabolic diseases such as diabetes mellitus.
6. Patients treated with anticoagulants, or using drugs that may affect visceral hemodynamics or portal pressure within the last 2 weeks.
7. Severe coagulation dysfunction, international normalized ratio > 5.
8. Those who are unable to lie flat or cannot tolerate the procedure.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study intended to include patients with hepatitis B cirrhosis who underwent HVPG examination in the hepatology outpatient/inpatient department as the case group, and healthy controls from the physical examination department, including 50 patients with HVPG <10 mmHg and 50 patients with HVPG ≥10 mmHg in the case group, and 50 healthy controls in the control group.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-09-14 (Estimated); Study Completion 2023-09-14 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the features of metabolomics for assessing portal hypertension in patients with hepatitis B cirrhosis | 12 months
  With HVPG as reference standard, the overall diagnostic performance (accuracy) for cirrhosis and portal hypertension of metabolomics was assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, M.D., Study Chair — Portal Hypertension Alliance in China; Ying Guo, M.D., Principal Investigator — The Third People's Hospital of Taiyuan; Jiaojian Lv, M.D., Principal Investigator — Lishui Country People's Hospital; Yang Wang, M.D., Principal Investigator — Shenyang Sixth People's Hospital; Shirong Liu, M.D., Principal Investigator — QuFu People's Hospital; Huadong Yan, M.D., Principal Investigator — Shulan (Hangzhou) Hospital
Locations (1):
- The Third People's Hospital of Taiyuan, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang X, Lin SX, Tao J, Wei XQ, Liu YT, Chen YM, Wu B. Study of liver cirrhosis over ten consecutive years in Southern China. World J Gastroenterol. 2014 Oct 7;20(37):13546-55. doi: 10.3748/wjg.v20.i37.13546. PMID 25309085
- [Background] Groszmann RJ, Wongcharatrawee S. The hepatic venous pressure gradient: anything worth doing should be done right. Hepatology. 2004 Feb;39(2):280-2. doi: 10.1002/hep.20062. No abstract available. PMID 14767976
- [Background] Abraldes JG, Sarlieve P, Tandon P. Measurement of portal pressure. Clin Liver Dis. 2014 Nov;18(4):779-92. doi: 10.1016/j.cld.2014.07.002. Epub 2014 Aug 21. PMID 25438283
- [Background] de Franchis R, Bosch J, Garcia-Tsao G, Reiberger T, Ripoll C; Baveno VII Faculty. Baveno VII - Renewing consensus in portal hypertension. J Hepatol. 2022 Apr;76(4):959-974. doi: 10.1016/j.jhep.2021.12.022. Epub 2021 Dec 30. PMID 35120736
- [Background] Zhang CE, Niu M, Li Q, Zhao YL, Ma ZJ, Xiong Y, Dong XP, Li RY, Feng WW, Dong Q, Ma X, Zhu Y, Zou ZS, Cao JL, Wang JB, Xiao XH. Urine metabolomics study on the liver injury in rats induced by raw and processed Polygonum multiflorum integrated with pattern recognition and pathways analysis. J Ethnopharmacol. 2016 Dec 24;194:299-306. doi: 10.1016/j.jep.2016.09.011. Epub 2016 Sep 9. PMID 27620661
- [Background] Wang X, Wang X, Xie G, Zhou M, Yu H, Lin Y, Du G, Luo G, Jia W, Liu P. Urinary metabolite variation is associated with pathological progression of the post-hepatitis B cirrhosis patients. J Proteome Res. 2012 Jul 6;11(7):3838-47. doi: 10.1021/pr300337s. Epub 2012 Jun 7. PMID 22624806